CLINICAL TRIAL: NCT03833271
Title: The Investigation of Immune Function and the Effectiveness of Influenza Vaccine in Children With Juvenile Idiopathic Arthritis Compared to Healthy Control
Brief Title: The Efficacy of Influenza Vaccine Program in Children With Juvenile Idiopathic Arthritis. A Single Centre Results From Hungary
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Nagy Arnold, Principal Investigator, University of Pecs
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MS Pecs-Paediatrics
Record Dates: First submitted 2019-01-21; First posted 2019-02-06 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Influenza Vaccines; Immune System Phenomena

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TNF-alpha inhibitor (Active Comparator)
  Interventions: Biological: Influenza vaccine, Immune function
- Methotrexate (Active Comparator)
  Interventions: Biological: Influenza vaccine, Immune function
- Healthy (Active Comparator)
  Interventions: Biological: Influenza vaccine, Immune function

INTERVENTIONS:
Biological: Influenza vaccine, Immune function — Comparing immune function and seroconversion after immunizing healthy children and juvenile idiopathic arthritis (JIA) children treated with different type of medication with influenza vaccine.

SUMMARY:
The aim of our study is to compare the immune function of patient treated with DMARD (methotrexate), or tumor necrosis factor (TNF)-alpha inhibitor (adalimumab) to healthy children. The study consists of three parts. In each part physical examination and routine laboratory tests are done.

At the first examination flow cytometry analysis is performed, after that the participants are immunized with influenza (3Fluart) vaccine. At part two and three further flow cytometry is carried out and seroconversion is measured.

ELIGIBILITY:
Inclusion Criteria:

* JIA (oligoarticular, polyarticular) treated with MTX or MTX/adalimumab
* Healthy controls

Exclusion Criteria:

* Children with infection
* Children with active JIA disease
* JIA other than oligoarticular, polyarticular type

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2018-10-28 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Comparing the healthy population and the JIA participants treated with DMARD (MTX) or TNF-alpha inhibitor (adalimumab) | 12-14 weeks
  Analysing T and B cells (%, /microL) by flow cytometry.
Immune response to influenza vaccine, the rate of seroconversion | 12-14 weeks
  Measuring seroconversion after influenza vaccine (IU)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pécs, Medical School, Department of Paediatrics, Pécs, Hungary

REFERENCES:
- [Derived] Nagy A, Mosdosi B, Simon D, Dergez T, Berki T. Peripheral Blood Lymphocyte Analysis in Oligo- and Polyarticular Juvenile Idiopathic Arthritis Patients Receiving Methotrexate or Adalimumab Therapy: A Cross-Sectional Study. Front Pediatr. 2020 Dec 10;8:614354. doi: 10.3389/fped.2020.614354. eCollection 2020. PMID 33363071